CLINICAL TRIAL: NCT04407403
Title: A Comparison of the Practice of Two Tai Chi Interventions Tailored for Different Health Outcomes
Brief Title: Health Outcomes of Two Different Tai Chi Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Linda Pescatello, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H16-262
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Fall
Keywords: Tai Chi; Hypertension; Balance function; Older adults
MeSH Terms: conditions — Hypertension | interventions — Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi tailored for lowering blood pressure (PRESSURE) (Experimental): During the 12-week Tai Chi intervention, participants in the PRESSURE group attended supervised Tai Chi sessions led by a certified Tai Chi instructor for 3 sessions/week, 60 minutes/session for 12 weeks. In addition, participants in the PRESSURE group were instructed: 1) to maintain their regular level of physical activity outside of the supervised Tai Chi exercise sessions, and diet during the study; and 2) to inform the researchers when there is a change(s) in a medical condition or medication prescribed.
  Interventions: Behavioral: Tai Chi tailored for lowering blood pressure (PRESSURE)
- Tai Chi tailored for improving balance (BALANCE) (Experimental): During the 12-week Tai Chi intervention, participants in the BALANCE group attended supervised Tai Chi sessions led by a certified Tai Chi instructor for 3 sessions/week, 60 minutes/session for 12 weeks. In addition, participants in the BALANCE group were instructed: 1) to maintain their regular level of physical activity outside of the supervised Tai Chi exercise sessions, and diet during the study; and 2) to inform the researchers when there is a change(s) in a medical condition or medication prescribed.
  Interventions: Behavioral: Tai Chi tailored for improving balance (BALANCE)
- control group (CONTROL) (No Intervention): During the 12-week Tai Chi intervention, participants in the CONTROL group performed their regular daily activities. In addition, participants in the CONTROL group were instructed: 1) to maintain their regular level of physical activity and diet during the study; and 2) to inform the researchers when there is a change(s) in a medical condition or medication prescribed. Of note, both PRESSURE and BALANCE were offered to participants assigned in the CONTROL group after data collection was completed.

INTERVENTIONS:
Behavioral: Tai Chi tailored for lowering blood pressure (PRESSURE) — PRESSURE Tai Chi routine consisted of eight forms following Yang style. PRESSURE was tailored for the targeted health outcome of BP in consultation with the professional, certified Tai Chi instructor and an experienced physical therapist. Specifically, investigators tailored PRESSURE to emphasize slow, deep breathing and relaxation by utilizing Tai Chi movements that: 1) were slow and smooth; 2) without break or pause; and 3) had minimal muscular force and exertion. Investigators included the following eight forms in PRESSURE: 1) Begin Tai Ji Quan; 2) Part the Horse's Mane; 3) Brush Knee and Push; 4) Cloud Hands; 5) Open and Close; 6) Part the Grass; 7) Single Whip; and 8) Finish Tai Ji Quan.
  Arms: Tai Chi tailored for lowering blood pressure (PRESSURE)
Behavioral: Tai Chi tailored for improving balance (BALANCE) — BALANCE Tai Chi routine consisted of eight forms following Yang style. BALANCE was tailored for the targeted health outcome of balance in consultation with the professional, certified Tai Chi instructor and an experienced physical therapist. Specifically, investigators tailored BALANCE to provide moderate to high levels of challenge to balance control by emphasizing movement principles (e.g., consciously control weight shifting during multi-directional stepping), and integrating Tai Chi movements that: 1) reduced the base of support; 2) moved the center of gravity; and 3) improved lower-extremity strength. Investigators included the following eight forms in BALANCE: 1) Begin Tai Ji Quan; 2) Roll the Ball; 3) Kick with Heel; 4) Repulse the Monkey; 5) Gather the Earth's Qi; 6) White Crane Spread Wing; 7) Fairy Weaves the Shuttle; and 8) Finish Tai Ji Quan.
  Arms: Tai Chi tailored for improving balance (BALANCE)

SUMMARY:
Tai Chi results in numerous health benefits but whether it can be tailored to elicit different health outcomes is not clear. Therefore, investigators compared the health benefits of two different Tai Chi interventions tailored for improvements in blood pressure (BP) (PRESSURE) or balance (BALANCE). Investigators tailored PRESSURE to emphasize breathing techniques and mental relaxation and BALANCE to emphasize movement principles that challenged balance. Participants were randomized to PRESSURE (n=12), BALANCE (n=13), or CONTROL (n=10). Tai Chi was practiced 3 sessions/week, 60 minute/session for 12 weeks. CONTROL performed normal daily activities. Investigators tested the change in cardiometabolic health, balance, and functional fitness outcomes among groups. Investigators hypothesized that PRESSURE would elicit greater BP reductions compared to BALANCE; meanwhile, BALANCE would elicit greater improvements in balance measures than PRESSURE.

DETAILED DESCRIPTION:
By 2030, older adults (≥65 years) will comprise approximately 20% (~72 million) of the United States (US) population. Currently in the US, over 70% of older adults have hypertension, and approximately 30% of healthy US older adults experience a fall annually. Therefore, preventing and treating high blood pressure (BP) and improving balance to reduce falling are priorities for healthy aging. Tai Chi is a low impact, social, and enjoyable form of exercise that is particularly suitable for older adults. In addition, BP and balance are the two most studied health outcomes of Tai Chi. Of note, Tai Chi varies considerably in terms of the styles (e.g., Yang), forms (e.g., cloud hands), and combinations of breathing techniques, mental relaxation, and movement principles. However, Tai Chi is rarely tailored for the health outcomes being targeted in research studies. Therefore, it is still unclear if healthcare professionals should recommend or design specific types of Tai Chi practice based on the health outcomes being targeted to maximize the benefits.

Investigators compared two different Tai Chi interventions, one tailored for reductions in BP (PRESSURE) and the other for improvements in balance (BALANCE) for their resultant health benefits among community dwelling older adults. Investigators hypothesized that PRESSURE would elicit statistically significantly greater BP reductions compared to BALANCE; meanwhile, BALANCE would elicit statistically significantly greater improvements in balance measures than PRESSURE.

All participants participated in three research visits. Visit1, and Visit 2 before, and Visit 3 after the 12-week Tai Chi exercise intervention or control group assignments. During Visit 1, investigators: 1) measured resting BP and completed the screening checklist; 2) administered questionnaires assessing life style habits (i.e., the Paffenbarger Physical Activity Questionnaire, the Block Rapid Food Screener, the Pittsburgh Sleep Quality Index), mental health (i.e., the Perceived Stress Scale Short Form, the Geriatric Anxiety Inventory); and 3) gave participants accelerometers to wear at home for 96 consecutive hours to measure habitual physical activity levels. Between Visits 1 and 2, investigators: 1) obtained medical clearance for all participants; and 2) perform the randomization of participants. During Visit 2, investigators assessed balance function (i.e., the Single Leg Stance Test, the Timed Up and Go Test, the Four Square Step Test, the Postural Stability Test, the Limits of Stability Test, the Modified Clinical Test of Sensory Interaction and Balance Test); BP; and functional fitness (i.e., the Hand Grip Test, the 30-Second Sit-to-Stand Test, the Chair Sit-and-Reach Test, the 10-Meter Walk Test). During the 12-week Tai Chi exercise intervention or control group assignments, participants assigned to BALANCE and PRESSURE groups were asked to attend Tai Chi exercise sessions for 3 sessions/week 60 minutes/session. Participants assigned to the control group did attend Tai Chi exercise sessions and were asked to maintain their regular level of physical activity. During Visit 3, investigators administered all measurements completed in Visit 2, and questionnaires administered in Visit 1.

ELIGIBILITY:
Inclusion Criteria:

1. The participant was enrolled in one of the three programs at Seabury including: the Seabury at Home program, the Independent Living program, and the Assisted Living program.
2. The participant was 50 or older, which was the age limit to be enrolled in any Seabury programs.
3. The participant was ambulatory without using an assistive device (e.g., walkers, canes, crutches).

Exclusion Criteria:

* 1. Older adults who enrolled in the Memory Support Assisted Living program or the Skilled Nursing program at Seabury were not invited to participate because Tai Chi practice could be too cognitively and/or physically challenging for them.

  2. To ensure the safety of exercise and avoid potential exercise-related cardiac events, if the participant had blood pressure (BP) be systolic BP <90 and/or systolic BP ≥160 mmHg and/or diastolic BP <60 and/or diastolic BP ≥100 mmHg during screening, this participant was excluded from further participation.

  3. Participants were removed from the study if they were not willing to comply with all study procedures. Participants were also removed from the study in the event of injury, illness, or other change that may influence the outcome variables being measured.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Resting Blood Pressure (BP) | Changes in resting SBP and DBP were calculated as the post-intervention resting BP measured at Visit 3 in week 14 minus the pre-intervention resting BP measured at Visit 2 in week 1.
  Investigators measured resting systolic BP (SBP) and resting diastolic BP (DBP) according to standards set by the American Heart Association using the OMRON automated BP monitors model HEM-705CPN in mmHg.
Change in the Single Leg Stance Test (SLS) | Changes SLS were calculated as the post-intervention SLS measured at Visit 3 in week 14 minus the pre-intervention SLS measured at Visit 2 in week 1.
  The SLS is a validated clinical test to measure static balance. Participants balanced on their dominant leg for as long as they can without any assistance from the ground or other objects. Investigators measured the seconds of successful balance using a handheld stopwatch.
Change in the Timed Up and Go Test (TUG) | Changes in TUG were calculated as the post-intervention TUG measured at Visit 3 in week 14 minus the pre-intervention TUG measured at Visit 2 in week 1.
  The TUG is a valid clinical test that was developed to assess dynamic balance and mobility in older adults. Following the word "Go", participants stood up from a standard chair (46 cm seat height, 65 cm armrest height), walk three meters as quickly as they could to a mark on the floor, turn and sit back down to the chair. Investigators measured the seconds used to finish the trial using a handheld stopwatch.
Change in the Four Square Step Test (FFS) | Changes in FFS were calculated as the post-intervention FFS measured at Visit 3 in week 14 minus the pre-intervention FFS measured at Visit 2 in week 1.
  The FFS is a validated dynamic standing balance test that puts high demand on the ability to plan and recall movements and execute those movements in a correct sequence. During the test, participants were asked to step in a predetermined sequence over four 90-cm-long walking sticks, placed in a cross configuration on the ground. The participant's starting position is in square 1 facing square 2. Then, the participant stepped forward, to the right, backward, and to the left into each quadrant in the clockwise direction, followed by the reverse sequence in the counterclockwise direction (i.e., the sequence 2, 3, 4, 1, 4, 3, 2, 1). Participants were instructed to complete the sequence as fast as possible without touching the sticks. Investigators measured the seconds used to finish the trial using a handheld stopwatch.
Change in the Postural Stability Test (PST) | Changes in PST were calculated as the post-intervention PST measured at Visit 3 in week 14 minus the pre-intervention PST measured at Visit 2 in week 1.
  The PST is a validated test to assess overall ability to maintain center of mass. It was administered using the Biodex Balance System SD (BBS) (Biodex Medical Systems, Shirley, USA). Investigators used the default setting that the stability of the platform was set on 8 (12 is the most stable, and 1 is the least stable). Participants stood on the platform with both feet and remain as still as possible. Each participant performed three 20-second trials, with ten seconds rest between trials. The BBS software (Biodex Medical Systems, Inc., version 1.3.4) calculated the medial-lateral stability index, the anterior-posterior stability index, and the overall stability index.
Change in the Limits of Stability Test (LST) | Changes in LST were calculated as the post-intervention LST measured at Visit 3 in week 14 minus the pre-intervention LST measured at Visit 2 in week 1.
  The LST is a validated test to assess functional stability limits, and anticipatory postural control. The LST was administered with the Biodex Balance System SD (BBS) (Biodex Medical Systems, Shirley, USA) following default settings. Reflecting the movement of the center of mass, a cursor on the screen in front of the participants were moved from a central circle to eight peripheral circles appearing successively in a random order on the screen. Participant were instructed to start moving the cursor toward the flashing target. The cursor had to stay within the target circle for a minimum of 0.5 seconds before it disappeared and showed the next target on the screen. Each trial ended when the eight target circles have been reached and the cursor repositioned in the central circle. The overall dynamic limit-of-stability score and the eight individual directional dynamic limit-of stability scores were calculated by the BBS software (Biodex Medical Systems, Inc., version 1.3.4).
Change in the Modified Clinical Test of Sensory Interaction and Balance (CTSIB) | Changes in CTSIB were calculated as the post-intervention CTSIB measured at Visit 3 in week 14 minus the pre-intervention CTSIB measured at Visit 2 in week 1.
  The CTSIB is a valid clinical assessment for investigating the sensory organization inputs in postural control. The CTSIB was administered with the Biodex Balance System SD (BBS) (Biodex Medical Systems, Shirley, USA) following default settings. Participants stood on the platform with both feet under four conditions: 1) eyes opened on firm surface; 2) eyes closed on firm surface; 3) eyes opened on a dynamic surface; and 4) eyes closed on dynamic surface. Each condition lasted 30 seconds with 10 seconds in between. A sway index was calculated for each of the four conditions by the BBS software (Biodex Medical Systems, Inc., version 1.3.4).

SECONDARY OUTCOMES:
Change in the Paffenbarger Physical Activity Questionnaire (PAFF) | Changes in PAFF were calculated as the post-intervention PAFF measured at Visit 3 in week 14 minus the pre-intervention PAFF measured at Visit 1 in week 1.
  The PAFF is a validated tool to assess habitual physical activity levels, including informal activities of daily living (e.g., city blocks walked, stairs climbed), leisure-time activities, and formal exercise. Activity scores in Kcal/week, and MET-minutes/week were calculated for walking, stair climbing, sport and leisure activity, and totaled. Activity scores in hours/week were calculated for sitting, light intensity, moderate intensity, and vigorous intensity activities.
Change in the Block Rapid Food Screener (BRFS) | Changes in BRFS were calculated as the post-intervention BRFS measured at Visit 3 in week 14 minus the pre-intervention BRFS measured at Visit 1 in week 1.
  The BRFS is a validated tool assess nutrient intake. It captures the nutrient intake such as dietary fat, and fiber, by collecting the frequency of consumptions of 24 food items (6 fruit/vegetable items, 3 bread/cereal items, and 15 meat/snack items). It was measured on a 5-point scale from 0 (Never, or less than once per week) to 4 (about 1 time per day or more).
Change in the Perceived Stress Scale Short Form (PSS) | Changes in PSS were calculated as the post-intervention PSS measured at Visit 3 in week 14 minus the pre-intervention PSS measured at Visit 1 in week 1.
  The PSS is a validated tool to assess the level of perceived stress. It assesses the extent to which situations during the past month have been perceived as stressful. It has 10 individual items which are measured on a 6-point scale from 0 (never) to 5 (very often).
Change in the Geriatric Anxiety Inventory (GAI) | Changes in GAI were calculated as the post-intervention GAI measured at Visit 3 in week 14 minus the pre-intervention GAI measured at Visit 1 in week 1.
  The GAI is validated tool to assess level of anxiety. It assesses typical common anxiety symptoms. The measurements of somatic symptoms with the instrument are limited in order to minimize confusion between symptoms common to anxiety and general medical conditions. This questionnaire has 20 individual questions that were answered as "agree" or "disagree".
Change in the Hand Grip Test (HGT) | Changes in HGT were calculated as the post-intervention HGT measured at Visit 3 in week 14 minus the pre-intervention HGT measured at Visit 2 in week 1.
  The HGT is a validated test as an indicator of overall body strength. The HGT was performed on the dominant arm with a calibrated Jamar Hydraulic Handgrip Dynamometer model 5030J1 (Lafayette Instrument Co., Lafayette, IN) in its second handle position. Participants were sitting with the arm against the trunk and the elbow flexed 90 degrees on the tested side.
Change in the 30-Second Sit-to-Stand Test (STS) | Changes in STS were calculated as the post-intervention STS measured at Visit 3 in week 14 minus the pre-intervention STS measured at Visit 2 in week 1.
  The STS is a validated test for assessing lower extremity strength. Participants were sitting in a standard padded chair (43.20 cm) without armrests and performed the test with both arms crossed against the chest. Participants started from the seated position, and then stood up until legs were straight and sat down with full weight placed on the chair. Investigators counted the number of chair stands completed in 30 seconds.
Change in the Chair Sit-and-Reach Test (CSRT) | Changes in CSRT were calculated as the post-intervention CSRT measured at Visit 3 in week 14 minus the pre-intervention CSRT measured at Visit 2 in week 1.
  The CSRT is a validated test for assessing hamstring flexibility. Participants sat in a chair with one leg extended and the other bent, then reached down and forward slowly in an attempt to touch the toes of the extended leg. Participants held a brief static position for 2 seconds, while investigators recorded the distance between the tips of the middle fingers and the middle of the toe at the end of the shoe in cm using an 18-inch (46 cm) ruler positioned parallel to the shin.
Change in the 10-Meter Walk Test (10MWT) | Changes in 10MWT were calculated as the post-intervention 10MWT measured at Visit 3 in week 14 minus the pre-intervention 10MWT measured at Visit 2 in week 1.
  : The 10-Meter Walk Test is a validated test for assessing participants' walking speed which is an important indicator of survival rates of older adults. Participants walked as fast as possible through a 15-meter walking path with 2.5 meters provided for acceleration and deceleration on each end. Investigators measured the seconds used to pass the data collection area at 10 meters with a handheld stopwatch. The fast walking speed (cm/second) was calculated for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Pescatello, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Seabury, Bloomfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No